CLINICAL TRIAL: NCT02324998
Title: A Study Into the Pharmacodynamic Biomarker Effects of Olaparib (a PARP Inhibitor) ± Degarelix (a GnRH Antagonist) Given Prior to Radical Prostatectomy
Brief Title: Study of Olaparib (± Degarelix) Given to Men With Intermediate/High Risk Prostate Cancer Before Prostatectomy
Acronym: CaNCaP03
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, CCTU- Cancer Theme, Cambridge Clinical Trials Unit - Cancer Theme, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CaNCaP03; 2014-004417-86 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: Radical Prostatectomy; Prostate Cancer; PARP inhibition; Olaparib; Degarelix; Neoadjuvant; Pharmacodynamics; Pharmacokinetics; Biomarkers
MeSH Terms: conditions — Prostatic Neoplasms | interventions — olaparib; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Olaparib Monotherapy
  Interventions: Drug: Olaparib
- Group B (Experimental): Olaparib in combination with degarelix
  Interventions: Drug: Olaparib; Drug: Degarelix

INTERVENTIONS:
Drug: Olaparib — PARP Inhibitor
  Other Names: AZD2281; Lynparza
Drug: Degarelix — Gonadotrophin releasing hormone blocker
  Other Names: Firmagon
  Arms: Group B

SUMMARY:
Despite recent advances in the treatment of Castrate-Resistant Prostate Cancer (CRPC), there remains an unmet medical need to identify and optimise additional treatment for those patients with early prostate cancer who are at greatest risk of relapse following first-line treatment with curative intent.

This is a phase I study investigating the feasibility and tolerability of a short course of neoadjuvant treatment with olaparib, either as a monotherapy or in combination with degarelix) given in the window-of-opportunity prior to radical prostatectomy in men with early, localised intermediate-/high- risk prostate cancer. Our primary objective is to determine the pharmacodynamic biomarker effects of olaparib (a PARP inhibitor) in this patient population.

Participants will receive either single agent olaparib or olaparib in combination with degarelix (androgen deprivation) for two weeks prior to routine radical prostatectomy. We will use immunohistochemistry to quantify changes in the levels of biomarkers of PARP inhibition, e.g. PAR, gamma H2AX, pH2A(s129) and Rad51 foci, using tumour samples taken at baseline and at the time of radical prostatectomy. An intra-operative prostate biopsy will permit us to examine biomarker variability between the samples.

The incidence and severity of Adverse Events will be documented and we will assess the number of trial participants who undergo surgery on schedule. We will assess preliminary evidence of tumour response, e.g. pathological changes and Prostate Specific Antigen (PSA). We also intend to investigate changes to the ctDNA profile by comparing blood samples collected throughout the study.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial the patient must:

* Have given written informed consent to participate*
* Men aged 18 years or over
* Patients suitable for radical prostatectomy
* ECOG performance status of 0 or 1
* Access to archived diagnostic tissue or consent to undergo repeat biopsy, if necessary
* Diagnosis of High risk or Intermediate risk prostate cancer, defined as:

  * High risk disease: one or more of stage T2c - 3a, or PSA level >20ng/mL, or Gleason score ≥ 8
  * Intermediate risk disease: two or more of: Stage T2 (any), PSA > 10, Gleason of ≥ 7
* Adequate bone marrow reserve and organ function (measured within 28 days prior to planned first olaparib administration) as demonstrated by the following values:

  * Absolute neutrophil count ≥ 1.8 x 109/L
  * Haemoglobin ≥ 117g/L
  * Platelet count ≥ 135 x 109/L
  * WBC ≥ 3.6 x 109/L
  * Peripheral blood smear with no features of MDS/AML
  * Adequate hepatic function:

    * Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of normal (ULN) AND
    * Total bilirubin ≤ 1.5 times the ULN unless in the presence of Gilbert's syndrome with an elevated indirect fraction
  * Adequate renal function:

    * Serum creatinine ≤ 1.5 times the ULN concurrent with creatinine clearance ≥ 50mL/min (calculated by Cockcroft and Gault equation)
* Willing to use two highly effective forms of contraception (see section 11.8) throughout their participation in the trial and for three months after their last dose of olaparib. Patients must refrain from donating sperm from the start of dosing up until sixteen weeks after discontinuing trial treatment
* Normal chest radiograph (CXR) and oxygen saturations
* Patients who are currently/have recently been involved in non-drug-based research are eligible to participate

  * If the patient does not consent to participate in the optional genetic research (ctDNA studies on blood) or to optional additional biopsies there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the trial.

Exclusion Criteria:

The presence of any of the following will preclude patient inclusion:

* Contraindication to olaparib or degarelix
* History of hypersensitivity to active or inactive excipients of olaparib
* Patients with known hypersensitivity to the degarelix active substance or mannitol must not receive degarelix.
* Current refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of olaparib
* As judged by the Investigator, any patient considered a poor medical risk due to a serious uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection including but not limited to:

  * Uncontrolled ventricular arrhythmia
  * Recent myocardial infarction (within three months)
  * Unstable spinal cord compression
  * Superior vena cava syndrome
  * Extensive bilateral lung disease on High Resolution Computed Tomography (HRCT)
  * History of pneumonitis
  * Active infection including hepatitis B, hepatitis C and Human Immunodeficiency Virus. Screening for chronic conditions is not required.
* Major surgery within 4 weeks prior to entry into the trial (excluding placement of vascular access). Patients must have recovered from side effects of any major surgery. Minor surgery (not including the diagnostic prostate biopsy) within 2 weeks prior to entry into the trial.
* Patients who have received (within last 3 months of trial entry) an investigational drug within a clinical trial will not be eligible to participate.
* Concomitant use of known potent CYP3A4 inhibitors and inducers. See section 10.4.1.1 for list and consider wash out periods.
* Blood transfusions within 1 month prior to the trial start
* ECG with mean resting QTc of ≥ 470ms (Fridericia; as per local reading) on two or more time points within a 24 hour period or family history of long QT syndrome
* Concomitant medications known to prolong the QT interval (see Appendix 1) or with factors that increase the risk of QTc prolongation or risk of arrhythmic events (such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age), History of Torsades de pointes.
* Judgement by the Investigator that the patient is unsuitable to participate in the trial and the patient is unlikely to comply with trial procedures, restrictions and requirements
* Patients with MDS or AML, or other previous malignancy except patients that have undergone treatment with curative intent for prior malignancy with no evidence of active prior malignancy are eligible.
* With the exception of alopecia, any unresolved toxicities from prior chemotherapy should be no greater than CTCAE (version 4.03) Grade 1 at the time of starting olaparib treatment.
* Patients with a desire to have children following the trial will not be recruited

Ages: 18 Years to 73 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-12; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Determination of PARP Inhibition | Two week olaparib therapy (alone or in combination with degarelix)
  Measure the degree of PARP inhibition by comparison of tumour samples taken from men with early prostate cancer at baseline and following treatment with olaparib (either alone or in combination with degarelix). Inhibition of PARP will be measured by the change in IHC levels of biomarkers such as PAR, gamma H2AX, pH2A(s129), Rad51 foci, FancD2 foci and ATM/ATR/CHK1/2.

SECONDARY OUTCOMES:
Incidence and Severity of Adverse Events | Two week olaparib therapy (alone or in combination with degarelix)
  Determine the incidence and severity of adverse events caused by treatment for 14 days with olaparib (either alone or in combination with degarelix) prior to radical prostatectomy. The severity of adverse events will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4.03).
Feasibility of treatment approach | Two week olaparib therapy (alone or in combination with degarelix)
  Assess the number of patients who undergo radical prostatectomy on schedule after 14 days of treatment with olaparib (either alone or in combination with degarelix).
Clinical benefit rate | Two week olaparib therapy (alone or in combination with degarelix)
  To assess preliminary evidence of tumour response, e.g. pathological changes and Prostrate Specific Antigen (PSA) levels, following 14 days treatment with olaparib (±degarelix).

OTHER OUTCOMES:
DNA repair defect and PARP inhibition | Two week olaparib therapy (alone or in combination with degarelix)
  Measure the DNA damage response, to compare with effects of or response to two weeks olaparib treatment (± degarelix)
Immunomodulatory effects of PARP inhibition | Two week olaparib therapy (alone or in combination with degarelix)
  Measure the immunophenotype, e.g. B and T cell subsets, of tumour samples taken at baseline and following 14 days treatment with olaparib (±degarelix) using, for example, IHC and FACS analysis.
Biological effects of PARP inhibition | Two week olaparib therapy (alone or in combination with degarelix)
  Measure biological effects, e.g. reduced tumour proliferation (Ki67), apoptosis (cleaved caspase 3) or altered androgen receptor/ETS regulated gene function in tumour samples taken from patients treated with olaparib.
Investigating changes to the ctDNA profile | Two week olaparib therapy (alone or in combination with degarelix)
  Measure changes in ctDNA profile following treatment with olaparib (either alone or in combination with degarelix).

CONTACTS AND LOCATIONS:
Overall Officials: Simon C Pacey, MRCP, Ph.D, Principal Investigator — University of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge University Hospitals Foundation Trust,, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No